CLINICAL TRIAL: NCT05979909
Title: Preventing Intravesical Recurrence in Patients With Urothelial Carcinoma of the Upper Urinary Tract: a Pilot Randomized Trial of a Single Prophylactic Bladder Instillation of Mitomycin C After Diagnostic Ureteroscopy
Brief Title: Intravesical Mitomycin C After Diagnostic Ureteroscopy for Upper Tract Urothelial Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14728
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Urothelial Carcinoma Ureter; Urothelial Cancer of Renal Pelvis
MeSH Terms: interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravesical mitomycin C (MMC) (Experimental)
  Interventions: Drug: Mitomycin C
- No intervention (No Intervention)

INTERVENTIONS:
Drug: Mitomycin C — Mitomycin (40 mg in 40 mL of sterile water) will be administered through a Foley catheter, which will be clamped for two hours.
  Arms: Intravesical mitomycin C (MMC)

SUMMARY:
The objective of this pilot study is to determine the feasibility of conducting a phase III randomized trial of intravesical mitomycin C (MMC) for prevention of intravesical recurrence (IVR) after diagnostic ureteroscopy for suspected upper tract urothelial carcinoma (UTUC). In the current study, 40 patients will be randomized to receive MMC or no intervention and will be followed for two years to determine the incidence of adverse events and IVR.

ELIGIBILITY:
Inclusion Criteria:

* Suspected upper tract urothelial carcinoma (UTUC)
* Diagnostic ureteroscopy required
* Tumor suggestive of upper tract urothelial carcinoma (UTUC) found on ureteroscopy

Exclusion Criteria:

* Prior or concomitant urothelial carcinoma of the bladder
* History of UTUC
* Ureteroscopy within the preceding six months
* Untreated urinary tract infection
* Suspected or confirmed perforation of the upper or lower urinary tract
* Lower urinary tract fistula
* Leukopenia or thrombocytopenia
* ECOG performance status 2 or greater
* Known hypersensitivity to mitomycin C
* Pregnancy or breastfeeding
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 30 days
  Proportion of patients who consent to participate in the study after being invited to do so
Randomization rate | 30 days
  Proportion of consented patients who are deemed eligible to participate and are randomly allocated to one of the two arms
Retention rate | 2 years
  Proportion of randomized patients who complete follow-up

SECONDARY OUTCOMES:
Adverse events (any) | 30 days
  Cumulative incidence of adverse events
Adverse events (severe) | 30 days
  Cumulative incidence of grade 3-5 adverse events
Intravesical recurrence | 2 years
  Cumulative incidence of urothelial carcinoma of the bladder

IPD SHARING:
Plan to Share IPD: No